CLINICAL TRIAL: NCT05254496
Title: Ensuring the Cultural Relevance of Dietary Guidelines Diet Patterns Among African Americans: Increasing Dietary Quality and Reducing Type 2 Diabetes Risk (Phase 2)
Brief Title: The Dietary Guidelines 3 Diet Patterns Study (DG3D): Phase 2
Acronym: DG3D-Phase2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00118661
Record Dates: First submitted 2022-02-23; First posted 2022-02-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to participant group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- US Healthy Diet (Experimental): Participants in this group will be assigned to follow the Healthy US dietary pattern as presented by the US Dietary Guidelines. As described here https://www.nia.nih.gov/health/usda-food-patterns: This eating pattern is based on the types and amounts of foods Americans typically consume. The main types of food in this eating pattern include a variety of vegetables; fruits; whole grains; fat-free or low-fat dairy; seafood, poultry, meat, and eggs; and nuts, seeds, and soy products.
  Interventions: Behavioral: Dietary Intervention Classes
- Mediterranean diet (Experimental): Participants in this group will be assigned to follow the Mediterranean dietary pattern as presented by the US Dietary Guidelines. As described here https://www.nia.nih.gov/health/usda-food-patterns: This eating pattern contains more fruits and seafood and less dairy than the Healthy U.S.-Style Eating Pattern.
  Interventions: Behavioral: Dietary Intervention Classes
- Vegetarian diet (Experimental): Participants in this group will be assigned to follow the Vegetarian dietary pattern as presented by the US Dietary Guidelines. As described here https://www.nia.nih.gov/health/usda-food-patterns: This eating pattern contains no meat, poultry, or seafood. Compared with the Healthy U.S.-Style Eating Pattern, it contains more soy products, eggs, beans and peas, nuts and seeds, and whole grains.
  Interventions: Behavioral: Dietary Intervention Classes

INTERVENTIONS:
Behavioral: Dietary Intervention Classes — Participants will attend classes once per week for 6 months and then bi-weekly for 6 months.

SUMMARY:
Based on the findings of our formative work, conduct a one-year intervention among African American Adults using revised culturally tailored materials to examine differences in Healthy Eating Index (HEI) and type 2 diabetes (T2DM) risk factors among participants (n=198) randomized to one of the 3 dietary patterns:

1) Healthy U.S.-Style Eating Pattern, 2) Healthy Mediterranean-Style Eating Pattern, and 3) Healthy Vegetarian Eating Pattern.

DETAILED DESCRIPTION:
The U.S. Dietary Guidelines (USDG) form the basis of federal nutrition programs and policy and provide valuable guidance to health initiatives and industries. The updated 2015 USDG moved away from a focus on individual nutrients to a greater focus on dietary patterns. The USDG state that healthy eating goals can be met through a variety of dietary patterns, but present healthy diet in three main ways: 1) Healthy U.S.-Style Eating Pattern, 2) Healthy Mediterranean-Style Eating Pattern, and 3) Healthy Vegetarian Eating Pattern. Currently, US adults are falling short of the nutrition recommendations (fruit/vegetable intake, greens/beans, whole grains, etc.) set forth by the USDG and measured by the Healthy Eating Index (HEI). While the USDG are the basis of nutrition guidelines, the research informing these dietary pattern recommendations has largely been drawn from observational studies among mostly white populations. In addition, there has been very limited cultural-tailoring of these dietary patterns that would ensure that these diets are acceptable to diverse populations, in particular, African Americans (AAs) living in the south, who experience a disproportionate burden of chronic disease, especially type 2 diabetes (T2DM). Currently, US adults are not meeting nutrition recommendations (fruit/vegetable, whole grains, etc.) set forth by the USDG and measured by the Healthy Eating Index (HEI).

For this study, AA adult participants with overweight/obesity and ≥three T2DM risk factors will be recruited to participate in the following aim:

Based on the findings of our formative work, conduct a one-year intervention using revised culturally tailored materials to examine differences in HEI and T2DM risk factors among participants (n=198) randomized to one of the 3 dietary patterns. This will result in community-based strategies around presenting dietary guidelines in a way to effectively meet nutrition recommendations leading to significant impacts on health among AA adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* BMI between 25- 49.9 kg/m2
* self-identify as African American
* live within 150 miles of the Columbia, SC area
* be able to attend all monitoring visits
* be willing to be randomized to one of the three conditions
* be free of major health or psychiatric diseases, drug or alcohol dependency, thyroid conditions, diabetes, or pregnancy

Exclusion Criteria:

* should not be pregnant (or have been pregnant in the last 6 months), anticipating on becoming pregnant in the next 12 months, or currently breastfeeding

  o Women who are pregnant should not be pursuing weight loss and should be under the direct care of a physician. Therefore women who are pregnant or who are anticipating they might be pregnant should not participate in this study. If a woman becomes pregnant during the study, she will be advised to consult with her healthcare provider and will be dropped from the weight loss study.
* should be free of an eating disorder as screened by the Eating disorder Screen for Primary care [ESP]. (If a participant has an eating disorder, they will be given contact information for the eating disorder clinic at the University of South Carolina)
* no current participation in a weight loss program or taking weight loss medications (although participants may be trying to lose weight on their own)
* no recent or planned bariatric surgery
* no recent weight loss (>10 lbs in the last 6 months)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in dietary quality | 12 months
  Changes in dietary quality as assessed by the Healthy Eating Index
Changes in body weight | 12 months
  Changes in body weight
Changes in HgbA1c | 12 months
  Changes in HgbA1c

SECONDARY OUTCOMES:
Changes in blood pressure | 12 months
  Changes in systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bailey S, Turner-McGrievy GM, Keseko EA, Duncan T, Ward-Johnson D, Davis B, Wilcox S, Friedman DB, Sarzynski MA, Liese AD. The Diet Guidelines: 3 Diets (DG3D) study protocol of a behavioral teaching kitchen intervention for type-2 diabetes prevention among African American adults. Contemp Clin Trials. 2025 Dec;159:108109. doi: 10.1016/j.cct.2025.108109. Epub 2025 Oct 10. PMID 41077220